CLINICAL TRIAL: NCT04419857
Title: A Randomized Control Trial to Determine Weight Gain Benefits of Caloric Supplementation for NAS Infants
Brief Title: A Trial to Determine Weight Gain Benefits of Caloric Supplementation for NAS Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028252; 2T35DK104689-06 (NIH)
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: high-caloric diet regimens
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-calorie formula (Experimental): Infant randomly assigned to high-calorie formula for 14 days
  Interventions: Dietary Supplement: High-calorie formula
- Standard calorie formula (No Intervention): Infant randomly assigned to standard-calorie formula for 14 days

INTERVENTIONS:
Dietary Supplement: High-calorie formula — Infant randomly assigned to high-calorie formula for 14 days
  Arms: High-calorie formula

SUMMARY:
A randomized clinical study in NAS infants managed via the Eat, Sleep, Console (ESC) approach comparing early weight loss on a standard-caloric density versus high-caloric density feeding regimen.

DETAILED DESCRIPTION:
The aims of the study is to systematically evaluate the benefit of high-caloric diet regimens given to NAS infants in the first three weeks of life. Breastfeeding is the preferred feeding method for NAS infants as it has shown to reduce NAS severity and infant weight loss, though women who are not adherent to drug treatment programs or have the potential to use illicit drugs are not able to breastfeed due to the risks posed to the infant. Several studies have demonstrated the potential for caloric enhancement of formula and breast milk to support weight gain in NAS infants. Through a randomized control trial analyzing infant weight gain on standard-calorie vs. high-calorie diet regimens, we aim to quantify weight patterns in NAS infants and show that increasing caloric intake can improve weight gain.

ELIGIBILITY:
Infant Inclusion Criteria:

* Infants with NAS born to mothers age 18-45 with methadone exposure before or during pregnancy who do not intend to place their infants for adoption
* Infants > 2200 g Infants at least 36 weeks gestational age
* Delivered at: Yale New Haven Hospital
* Mothers/infants able to return to outpatient pediatric provider for 2 month and 4 month weights visits

Infant Exclusion Criteria:

* Infants with major congenital malformations
* Infants enrolled to NICU >24 hours for medical conditions other than NAS treatment before 3 days of life

Mother's Inclusion criteria -

* Pregnant women (age 18-45) who have started methadone treatment at obstetrics or other YNHH appointments
* Confirm methadone treatment is received from a licensed treatment program
* Confirm that mothers are planning to deliver their infant(s) at Yale New Haven Hospital
* Confirm that mothers do not intend to place the infant(s) for adoption
* Confirm mother's willingness to participate in the study (including attending the 2-month and 4-month follow up weigh-ins with pediatrician)
* Consent forms will be signed and faxed to study staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Maximal percent weight loss compared to birth weight | 2 weeks
  this will be measured by twice daily weights while in the hospital and once daily weights at home for two weeks after birth compared with birth weight

SECONDARY OUTCOMES:
Hours to weight nadir | 2 weeks
  Measured by determining the hours of life that the maximal percent weight loss was obtained for each patient, assessed within the first two weeks after birth
Days to return to birthweight | 1 month
  Measured by determining the days of life each patient regained birthweight, assessed within the first month after birth
Percent weight change per day | 2 weeks
  Measured by comparing the weight from the weight obtained the day prior, assessed daily for the first two weeks after birth
Length of hospital stay | up to 6.5 days
  Measured by comparing admission time to discharge time, assessed at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Grossman, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No